CLINICAL TRIAL: NCT06609525
Title: A Multi-center, Double-blind, Randomized, Parallel, Active-controlled, Non-inferior, Phase Ⅱb/Ⅲ Study to Evaluate the Safety and Efficacy of CTO0303
Brief Title: Comparing Efficacy and Safety of CTO0303 in Pediatric Subjects
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CTO0303
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-01

CONDITIONS: Pupillary Dilation Effect During Cycloplegic Refraction
Keywords: pupillary dilation
MeSH Terms: conditions — Mydriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CTO0303-A (Experimental)
  Interventions: Drug: CTO0303-A
- CTO0303-B (Experimental)
  Interventions: Drug: CTO0303-B
- CTO0303-C (Active Comparator)
  Interventions: Drug: CTO0303-C

INTERVENTIONS:
Drug: CTO0303-A — eye drop, 1 drop 3 times (every 5 minutes) a day
  Arms: CTO0303-A
Drug: CTO0303-B — eye drop, 1 drop 3 times (every 5 minutes) a day
  Arms: CTO0303-B
Drug: CTO0303-C — eye drop, 1 drop 3 times (every 5 minutes) a day
  Arms: CTO0303-C

SUMMARY:
This is a prospective randomized study compared with active control arm.

DETAILED DESCRIPTION:
This is a prospective randomized study compared with active control arm. The investigators compare the pupil size in subject when 30 minutes after administering IP (CTO0303 or active control).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric or adolescent subjects those who get a written consent both whom and their parents (or legally acceptable representative)
* Pediatric or adolescent subjects aged 4 to 15 years old based on date of written consent

Exclusion Criteria:

* Subjects with a history of severe systemic reaction or increased sensitivity to atropine
* Subjects with anterior segment disease that interferes with ophthalmological examination (ex. corneal scar, corneal opacity and others)
* Subjects administered mydriatic medication within 14 days prior to administration of Investigational Product
* Subjects with contact lens

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
pupillary dilation effect at 30 minutes after administration | From enrollment to the end of treatment at 1 day.
  The pupil size is measured using a pupillometer 30 minutes after IP administration

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No